CLINICAL TRIAL: NCT04521595
Title: Expansion of the Weigh Smart Pediatric Group Family Oriented Weight Management Program Through the Use of Telehealth
Acronym: Weigh Smart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00251530
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- weigh smart intervention (Experimental): open treatment arm to receive group based lifestyle intervention via telehealth.
  Interventions: Behavioral: Weigh Smart Telehealth intervention

INTERVENTIONS:
Behavioral: Weigh Smart Telehealth intervention — Trial of the group program (nutrition, exercise) delivered via telehealth through fruit street on the Eastern Shore and Western Maryland with use of noninvasive lifestyle tracking options (drink water aquarium app for water consumption and fitbit - steps, sleep monitoring) provides novel options for expansion of family- based lifestyle intervention to underserved areas. We plan as a pilot study to assess the sensitivity of noninvasive measures for the detection of sleep apnea (pediatric sleep questionnaire (PSQ) and fitbit sleep data) in comparison to clinically indicated polysomnography among children with clinical suspicion for sleep apnea.

SUMMARY:
There has been a steep rise in the prevalence of obesity among children and adults in the United States. The Weigh Smart program, a family based weight management program was developed in 2005 with significant improvement in the severity of obesity among children in the Baltimore are participating in the group program with limited impact outside the region due to transportation. Trial of the group program (nutrition, exercise) delivered via telehealth through fruit street on the Eastern Shore and Western Maryland with use of noninvasive lifestyle tracking options (drink water aquarium app for water consumption and fitbit- steps, sleep monitoring) provides novel options for expansion of family- based lifestyle intervention to underserved areas. Investigators plan as a pilot study to assess the sensitivity of noninvasive measures for the detection of sleep apnea (pediatric sleep questionnaire (PSQ) and fitbit re: sleep data) in comparison to clinically indicated polysomnography among children with clinical suspicion for sleep apnea.

DETAILED DESCRIPTION:
. Trial of the group program (nutrition, exercise) delivered via telehealth through fruit street to families of overweight and obese children between 7-17 years of age referred from selected pediatric practices on the Eastern Shore of Maryland and Western Maryland with use of noninvasive lifestyle tracking options (drink water aquarium app for water consumption and fitbit charge 3- steps, sleep monitoring) provides novel options for expansion of family- based lifestyle intervention to underserved areas. Investigators plan as a pilot study to assess the sensitivity of noninvasive measures for the detection of sleep apnea (pediatric sleep questionnaire (PSQ) and fitbit charge 3 sleep data) in comparison to clinically indicated polysomnography among children with clinical suspicion for sleep apnea.

ELIGIBILITY:
Inclusion Criteria

* Children who are overweight/obese (7-17 years of age)
* Children must be referred by selected Maryland Eastern Shore and Western Maryland pediatric practices to Mount Washington Pediatric Hospital Weigh Smart. Families must provide informed consent at the weigh smart visit and have access to either a tablet, laptop or smart phone device to participate.

Exclusion Criteria

* Children outside of the age range
* Children not seen by Maryland Eastern Shore or Western Maryland pediatric providers who are part of the intervention group
* Children who do not have internet access either by smart phone or tablet to allow telehealth participation
* Children who are unwilling to participate in group program and followup local visits

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Combined Weight change in parent and child | Up to 12 months
  Comparison of combined weight of both child and parent at baseline to weight at 1,3,6 months post-intervention

SECONDARY OUTCOMES:
Change in Pediatric Sleep Questionnaire (PSQ) sleep questionnaire in child | up to 12 months
  This will assess the comparison of score at baseline to 3-6 months post-intervention. The PSQ contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric Obstructive Sleep Apnea features. It is a binary scale of 2 responses, YES=1 OR NO=0, therefore a maximum of 22 points and minimum of zero.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Washington Pediatric Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pilot study at present. Plan to present results once completed